CLINICAL TRIAL: NCT07239505
Title: The Role Of Trinase In Reducing Post-Operative Pain For Patients With Symptomatic Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: A Randomized Controlled Trial Evaluating Whether Pre-operative Trinase Reduces Post-operative Pain in Patients With Symptomatic Irreversible Pulpitis Compared to Placebo, Using VAS Scores and Analgesic Intake Over 48 Hours.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Sara Elmallah, Associate professor of Endodontics, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 102517
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Symptomatic Irreversible Pulpitis (SIP); Postoperative Pain After Endodontic Treatment; Endodontic Disease; Dental Pain
Keywords: Visual Analogue Scale (VAS); Randomized Controlled Trial; Trinase; Postoperative Pain
MeSH Terms: conditions — Dental Pulp Diseases; Toothache; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants are randomized into two parallel groups: Trinase vs. placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both participants and the treating clinician are blinded to allocation. Medication and placebo are packed in identical opaque envelopes prepared by an independent assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trinase group (Experimental): Patients receive one tablet of Trinase (trypsin, bromelain, and rutin) orally 30 minutes before single-visit root canal treatment (RCT). RCT is performed under local anesthesia (2% mepivacaine with 1:100,000 epinephrine), rubber dam isolation, using ProTaper Next rotary files up to X3, 2.5% NaOCl irrigation, EDTA gel, obturation with modified single-cone technique and Adseal resin sealer. Post-operative pain assessed via VAS at 6, 12, 24, 48 hours. Analgesic rescue (Trinase) allowed if needed; consumption recorded.
  Interventions: Drug: Trinase
- Placebo group (Placebo Comparator): Patients receive one identical-appearing placebo tablet orally 30 minutes before identical single-visit RCT procedure (same anesthesia, instrumentation, irrigation, obturation protocol). Post-operative pain assessed via VAS at 6, 12, 24, 48 hours. Analgesic rescue (Trinase) allowed if needed; consumption recorded.
  Interventions: Drug: placebo capsule

INTERVENTIONS:
Drug: Trinase — One tablet of Trinase (proteolytic enzyme combination: trypsin, bromelain, and rutin) administered orally 30 minutes prior to root canal treatment. Used as premedication to reduce postoperative pain and inflammation.
  Arms: Trinase group
Drug: placebo capsule — One identical-appearing placebo tablet administered orally 30 minutes prior to root canal treatment. Used as control.
  Arms: Placebo group

SUMMARY:
This study aims to determine whether Trinase, an enzyme-based anti-inflammatory medication, can reduce pain after root canal treatment in patients with symptomatic irreversible pulpitis. A total of 182 male patients aged 18 to 50 years who present with moderate to severe tooth pain will be randomly assigned to receive either a Trinase tablet or a placebo 30 minutes before treatment. All root canal procedures will be performed in a single visit using standard endodontic techniques.

Pain levels will be measured on a Visual Analogue Scale (VAS) before treatment and at 6, 12, 24, and 48 hours after treatment. Patients will also record the number of pain-relief tablets they take during the first 48 hours. The goal of the study is to see whether Trinase can lower post-operative pain and reduce the need for analgesic medication compared with placebo. This information may help improve pain management for patients undergoing root canal therapy.

DETAILED DESCRIPTION:
Symptomatic irreversible pulpitis is a common endodontic condition characterized by severe inflammatory dental pain. Although root canal treatment (RCT) is effective in removing the inflamed pulp tissue, many patients continue to experience pain during the first 24-48 hours after treatment. Post-operative endodontic pain affects patient comfort, satisfaction, and clinical workflow, making pain control an essential component of evidence-based endodontic care.

Traditional pharmacological methods for managing post-operative dental pain include nonsteroidal anti-inflammatory drugs (NSAIDs) and corticosteroids. While these medications are effective, they are also associated with potential gastrointestinal and systemic adverse effects, especially when used repeatedly. As a result, there is growing interest in alternatives that can reduce inflammation and discomfort while minimizing systemic risks. Enzyme-based anti-inflammatory therapies, including combinations of trypsin, bromelain, and rutin, have been shown in medical and dental literature to provide meaningful reductions in pain, edema, and inflammation following surgical procedures. These proteolytic enzymes act by breaking down inflammatory mediators, reducing tissue permeability, and modulating cytokine responses. Trinase, a formulation containing trypsin, bromelain, and rutin, is widely used in postoperative care in other medical fields, yet its role in managing pain following endodontic procedures has not been adequately studied.

This randomized, double-blind, placebo-controlled clinical trial is designed to evaluate whether administering Trinase before root canal treatment can reduce the intensity of post-operative pain in patients diagnosed with symptomatic irreversible pulpitis. A total of 182 systemically healthy male patients, aged 18 to 50 years, will be recruited from the Endodontics Department at Fayoum University. The study population is limited to male participants to standardize biological pain variability and hormonal influences on pain perception. Eligible patients must present with restorable mandibular molar teeth and moderate to severe preoperative pain confirmed both clinically and radiographically.

Participants will be randomly assigned to one of two equal study arms. The Trinase group will receive a single oral Trinase tablet 30 minutes before treatment. The placebo group will receive a visually identical tablet administered under the same conditions. An assistant not involved in treatment will prepare and code all medication envelopes, ensuring allocation concealment. Both the operator and the participants will be blinded to group assignment.

All treatments will be performed in a single visit using standardized endodontic procedures. After local anesthesia, rubber-dam isolation, and access preparation, canal patency will be confirmed using stainless steel hand files. Working length will be determined electronically and confirmed radiographically. Mechanical instrumentation will be performed using Protaper Next rotary instruments according to manufacturer instructions. Irrigation will be performed using 2.5% sodium hypochlorite and EDTA gel lubricant. Upon completion of cleaning and shaping, canals will be dried, obturated using a modified single-cone technique with resin-based sealer, and restored temporarily with intermediate restorative material. All procedures are performed by a single experienced operator to eliminate inter-operator variability.

The primary outcome measure is postoperative pain intensity assessed using a 10-cm Visual Analogue Scale (VAS). Patients will record their pain levels at baseline and at 6, 12, 24, and 48 hours after treatment. Pain will be categorized using validated VAS cutoff values. The secondary outcome measure is the total number of analgesic tablets consumed within 48 hours following treatment. Participants will receive a standardized pain diary to document both pain levels and analgesic intake.

Statistical analysis will be conducted using non-parametric tests due to expected non-normal distribution of pain scores. Between-group differences will be analyzed using the Mann-Whitney test, and within-group comparisons across time points will be performed using the Friedman test followed by appropriate post-hoc analysis. The significance level will be set at p ≤ 0.05. Sample size was calculated using PS software to detect clinically relevant differences in postoperative pain with an anticipated dropout rate accounted for by enrolling 182 participants.

The study protocol has been reviewed and approved by the Fayoum University Supreme Committee for Scientific Research Ethics (FU-SCSRE). Written informed consent will be obtained from each participant. The study involves minimal risk, as Trinase is a commercially available medication with a well-established safety profile and the placebo carries no known risks. The duration of active participation for each subject is approximately 48 hours, corresponding to the postoperative observation period. No additional radiographs or invasive procedures beyond standard clinical care will be performed.

This study aims to determine whether Trinase can serve as a simple, safe, and effective adjunct to improve postoperative patient comfort following root canal therapy. The results may help clarify the role of enzyme-based anti-inflammatory medications in endodontic pain management and potentially reduce reliance on traditional analgesics with known adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy male patients (ASA I or II)
* Aged 18 to 50 years
* Presenting with symptomatic irreversible pulpitis in a restorable mandibular molar
* Preoperative moderate to severe pain (VAS ≥45 mm)
* Normal periapical tissue (no radiolucency, pocket depth ≤5 mm, mobility ≤ Grade I)

Exclusion Criteria:

Medically compromised patients (ASA III or higher)

* History of allergy or intolerance to Trinase or any of its components (trypsin, bromelain, rutin)
* Vertical root fracture
* External or internal root resorption
* Periodontal pocket depth >5 mm
* Tooth mobility Grade II or III
* Presence of periapical lesion (radiolucency)
* Female patients (to standardize pain perception and hormonal factors)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain intensity assessed by Visual Analogue Scale (VAS) | 6, 12, 24, and 48 hours after root canal treatment
  Pain intensity recorded by patients on a 10-cm Visual Analogue Scale (VAS) where 0 = no pain and 100 = pain as bad as it could be. Scores categorized as: no pain (0-4 mm), mild (5-44 mm), moderate (45-74 mm), severe (75-100 mm). Measured at baseline and post-operatively.

SECONDARY OUTCOMES:
Number of analgesic tablets consumed within 48 hours post-treatment | Within 48 hours post-treatment
  Total number of rescue analgesic tablets (Trinase) taken by patients within 48 hours after root canal treatment, as recorded on provided charts during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) including demographics, baseline VAS, postoperative VAS scores (6, 12, 24, 48h), and analgesic consumption will be shared. Data will be anonymized (no names, IDs, or dates) and provided in CSV/SPSS format. IPD will be available 6 months after publication of primary results and for 5 years thereafter. Access requires a signed data use agreement specifying research purpose and ethics approval. Contact: Dr. Sara Samir Elmallah (sara.elmallah@fayoum.edu.eg).
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- See also: Description: Official ClinicalTrials.gov record for this study (NCT number assigned upon submission) — https://clinicaltrials.gov/study/NCT_TO_BE_ASSIGNED